CLINICAL TRIAL: NCT00232271
Title: The Effect of Enoxaparin Sodium (Clexane) on the Incidence of Deep Vein Thrombosis Following Electrophysiology Studies and Radiofrequency Ablation.
Brief Title: The Effect of Enoxaparin Sodium on the Incidence of Deep Vein Thrombosis Following Electrophysiology Studies and Radiofrequency Ablation.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Melbourne Health (Other)
Collaborators: Sanofi (Industry); National Heart Foundation, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2004-157
Record Dates: First submitted 2005-10-02; First posted 2005-10-04 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2005-10

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Enoxaparin

ARMS (2):
- clexane (Active Comparator): patients received clexane
  Interventions: Drug: Clexane
- non clexane (No Intervention): no clexane given

INTERVENTIONS:
Drug: Clexane
  Arms: clexane

SUMMARY:
The purpose of this study is to assess the effect of the anticoagulant(blood thinner) Clexane on the development of leg clots following electrophysiology studies (EPS) and or radiofrequency ablation (RFA).

People who suffer heart palpitations will sometimes need hospital admission to undergo an electrophysiology study ( and or a Radiofrequency Ablation)in order to diagnose and or treat their condition.

Radiofrequency ablation is a procedure to stop abnormal heart rhythms. EPS/RFA studies require the puncture of the leg veins . Previous experience has shown that following the puncture of leg veins there is a small risk of developing a blood clot in the leg.

It is not known whether giving blood thinners (anticoagulants) after the procedure will decrease this risk Enoxaparin Sodium (Clexane) is an anticoagulant used extensively and safely following bone (Orthopaedic) surgery to prevent blood clots from developing in the legs

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing EPS/RFA for the diagnosis and or treatment of SVT based on patient history or ECG evidence.

Exclusion Criteria:

* Patients with a past history of DVT or PE.
* Patients with a history of clotting disorders
* Patients with active malignancies
* Patients requiring full heparinisation during and after the procedure.
* Chronic atrial flutter and atrial fibrillation ablation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-08; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Incidence of deep vein thrombosis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sparks, MBBS, PhD. FRACP, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne hospital, Melbourne, Victoria, Australia